CLINICAL TRIAL: NCT02191579
Title: A Multicenter, Prospective, Randomized, Open-label Study to Compare the Efficacy, Safety, and Tolerability of BOTOX® and Topiramate for Headache Prophylaxis in Adults With Chronic Migraine
Brief Title: Efficacy and Safety Study of BOTOX® Compared to Topiramate for the Prevention of Chronic Migraine in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GMA-US-NEU-0206; FORWARD (Other: Allergan)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BOTOX® (Active Comparator): 155U onabotulinumtoxinA (BOTOX®) total dose per treatment by intramuscular injection every 12 weeks for up to 3 treatments.
  Interventions: Biological: onabotulinumtoxinA
- Topiramate (Active Comparator): Topiramate starting at a daily oral dose of 25 mg/day titrated up to a maximum dose of 100 mg/day for 36 weeks. Participants who discontinue topiramate are eligible to receive treatment with BOTOX®.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Biological: onabotulinumtoxinA — 155U onabotulinumtoxinA (BOTOX®) total dose per treatment by intramuscular injection every 12 weeks.
  Other Names: BOTOX®; botulinum toxin Type A
  Arms: BOTOX®
Drug: Topiramate — Topiramate up to a maximum oral dose of 100 mg/day.
  Other Names: Topamax®
  Arms: Topiramate

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of prophylactic (preventative) treatment with BOTOX® (onabotulinumtoxinA) compared to topiramate in adults with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic migraine
* More than 15 headache days in a 28 day period (headaches that last more than 4 hours and/or require treatment with prescription medication).

Exclusion Criteria:

* Taking opioid-containing products for acute headache treatment more than 8 days during a 28-day period
* Previous treatment with botulinum toxin of any serotype for any reason
* Previous treatment with topiramate
* On a ketogenic diet (high in fat, low in carbohydrates)
* History of acute myopia or increased intraocular pressure
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis or any other significant disease that might interfere with neuromuscular function
* Acupuncture, transcutaneous electrical stimulation (TENS), cranial traction, dental splints for headache, or injection of anesthetics/steroids in the 4 weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Jo, Study Director — Allergan
Locations (32):
- United States (32):
  - St Joseph's Hospital Barrow Neurology Clinics, Phoenix, Arizona
  - North County Neurology Associates, Encinitas, California
  - California Headache and Balance Center, Fresno, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Denver Neurological Clinic, Denver, Colorado
  - Ki Health Partners LLC DBA New England Institute for Neurology and Headache, Stamford, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton Inc, Boca Raton, Florida
  - Design Neuroscience Center, Doral, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Negroski, Sutherland & Hanes Neurology, Sarasota, Florida
  - Neurology Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Robbins Headache Clinic, Riverwoods, Illinois
  - International Clinical Research Institute Inc, Overland Park, Kansas
  - Kansas City Bone and Joint Clinic, Overland Park, Kansas
  - The NeuroMedical Center, Baton Rouge, Louisiana
  - MedVadis Research Corporation, Watertown, Massachusetts
  - New England Regional Headache Center Inc, Worcester, Massachusetts
  - Allegiance Health, Jackson, Michigan
  - Clinvest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Renown Institute for Neurosciences, Reno, Nevada
  - Dent Neurosciences Research Center Incorporated, Amherst, New York
  - Island Neurological Associates PC, Plainview, New York
  - Montefiore Headache Center, The Bronx, New York
  - Asheville Neurology Specialists PA, Asheville, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
  - Raleigh Neurology Associates PA, Raleigh, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Main Line Health Lankenau Hospital, Wynnewood, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - Puget Sound Neurology, Tacoma, Washington

REFERENCES:
- [Derived] Blumenfeld AM, Patel AT, Turner IM, Mullin KB, Manack Adams A, Rothrock JF. Patient-Reported Outcomes from a 1-Year, Real-World, Head-to-Head Comparison of OnabotulinumtoxinA and Topiramate for Headache Prevention in Adults With Chronic Migraine. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720959936. doi: 10.1177/2150132720959936. PMID 32985341
- [Derived] Rothrock JF, Adams AM, Lipton RB, Silberstein SD, Jo E, Zhao X, Blumenfeld AM; FORWARD Study investigative group. FORWARD Study: Evaluating the Comparative Effectiveness of OnabotulinumtoxinA and Topiramate for Headache Prevention in Adults With Chronic Migraine. Headache. 2019 Nov;59(10):1700-1713. doi: 10.1111/head.13653. Epub 2019 Sep 26. PMID 31559634

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate/BOTOX®: Topiramate starting at a daily oral dose of 25 mg/day titrated up to a maximum dose of 100 mg/day for 36 weeks. Participants who discontinue topiramate are eligible to receive treatment with BOTOX®.
Period: Treatment 1
Arm/Group | BOTOX® | Topiramate/BOTOX®
Started | 140 | 142
Completed | 113 | 84
Not Completed | 27 | 58
Not completed — Multiple Reasons Specified | 27 | 58
Period: Treatment 2
Arm/Group | BOTOX® | Topiramate/BOTOX®
Started | 0 | 80
Completed | 0 | 55
Not Completed | 0 | 25
Not completed — Multiple Reasons Specified | 0 | 25

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® | Topiramate | Total
Number analyzed (Participants) | 140 | 142 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.7) | 39.4 (12.6) | 39.8 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  18 to <25 | 16 | 21 | 37
  25 to <35 | 30 | 40 | 70
  35 to <45 | 43 | 29 | 72
  45 to <55 | 33 | 34 | 67
  ≥55 | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 122 | 239
  Male | 23 | 20 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 111 | 118 | 229
  Black | 13 | 8 | 21
  Asian | 4 | 2 | 6
  Hispanic | 11 | 12 | 23
  Other | 1 | 2 | 3
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 167.4 (8.5) | 167.0 (8.7) | 167.2 (8.5)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 81.0 (21.8) | 80.5 (20.6) | 80.8 (21.1)
Body Mass Index (BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (7.1) | 28.8 (6.5) | 28.8 (6.8)
Use of Headache Prophylactic Treatment(s) [Count of Participants; unit: Participants] | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 50% Decrease From Baseline in the Frequency of Headache Days
Description: Participants recorded their headaches in a daily e-diary. A headache day was defined as a calendar day (00:00 to 23:59) with 4 or more hours of headache and/or headache of any duration with the use of migraine-specific acute headache medication(s). The number of headache days over the 28-day period was counted. The percentage of participants with a ≥ 50% decrease in headache days in the 28-day period prior to Week 32 relative to Baseline (28-day period prior to Day 1) is reported.
Time Frame: Baseline (First 28 days from Screening) to the last 28-day period ending with Week 32
Population: ITT Set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX® | Topiramate
Number analyzed (Participants) | 140 | 142
percentage of participants | 40.0 | 12.0
Statistical Analysis 1: Comparison: BOTOX® vs Topiramate; Test type: Superiority; p < 0.001, Regression, Logistic — Odds ratio, 95% CI, and p-value were estimated using a logistic regression model adjusted by baseline headache days; Odds Ratio (OR) = 4.94, 95% CI 2-sided [2.681 to 9.085]

2. Secondary Outcome: Change From Baseline in the Frequency of Headache Days Per 28-day Period
Description: Participants recorded their headaches in a daily e-diary. A headache day was defined as a calendar day (00:00 to 23:59) with 4 or more hours of headache and/or headache of any duration with the use of migraine-specific acute headache medication(s). The number of headache days over the 28-day period was counted. A negative change from Baseline (less headache days) indicates improvement.
Time Frame: Baseline (First 28 days from Screening) to the last 28-day period ending with Week 32
Population: ITT Set included all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BOTOX® | Topiramate
Number analyzed (Participants) | 140 | 142
days | -8.3 (8.9) | -2.1 (5.6)
Statistical Analysis 1: Comparison: BOTOX® vs Topiramate; Test type: Superiority; p < 0.001, ANCOVA — Estimated mean difference, 95% CI, and p-value were assessed using analysis of covariance adjusting for baseline headache days; Mean Difference (Net) = -6.199, 95% CI 2-sided [-7.936 to -4.462]

3. Secondary Outcome: Change From Baseline in Headache Impact Test (HIT-6) Total Score
Description: The HIT-6 is a valid disease-targeted measure used to assess the impact of headaches, comprised of 6 items that assess pain, role functioning, social functioning, cognitive functioning, vitality, and psychological distress. A total score is created by summingacross all items, and ranges from 36 (no impact) to 78 (severe impact) reflecting a "best to worst" scoring.
  A negative change from Baseline (a lower score) indicates improvement.
Time Frame: Baseline (Day 1) to the last 28-day period ending with Week 30
Population: Participants from the ITT Set, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BOTOX® | Topiramate
Number analyzed (Participants) | 110 | 115
score on a scale | -5.6 (7.2) | -1.3 (3.9)
Statistical Analysis 1: Comparison: BOTOX® vs Topiramate; Test type: Superiority; p < 0.001, ANCOVA — Estimated mean difference, 95% CI, and p-value for Week 30 were assessed using analysis of covariance adjusting for baseline headache days; Median Difference (Net) = -4.248, 95% CI [-5.766 to -2.731]

4. Secondary Outcome: Percentage of Participants With a ≥ 70% Decrease From Baseline in the Frequency of Headache Days
Description: Participants recorded their headaches in a daily e-diary. A headache day was defined as a calendar day (00:00 to 23:59) with 4 or more hours of headache and/or headache of any duration with the use of migraine-specific acute headache medication(s). The number of headache days over the 28-day period was counted. The percentage of participants with a ≥ 70% decrease in headache days in the 28-day period prior to Week 32 relative to Baseline (28-day period prior to Day 1) is reported.
Time Frame: Baseline (First 28 days from Screening) to the last 28-day period ending with Week 32
Population: ITT Set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX® | Topiramate
Number analyzed (Participants) | 140 | 142
percentage of participants | 27.1 | 8.5
Statistical Analysis 1: Comparison: BOTOX® vs Topiramate; Test type: Superiority; p < 0.001, Regression, Logistic — Odds ratio, 95% CI, and p-value for the Week 29-32 interval were estimated using a logistic regression model adjusted by baseline headache days; Odds Ratio (OR) = 4.05, 95% CI [2.014 to 8.157]

ADVERSE EVENTS:
Time Frame: First dose of study drug to the final visit (Up to 48 Weeks)
Description: Adverse Events (AEs) were counted in the treatment group based on investigator's determination. If investigators determined AE was related to both treatments or relatedness was unknown, it was counted in both treatment groups, but only once for the total population.
Groups:
- BOTOX®: 155U onabotulinumtoxinA (BOTOX®) total dose per treatment by intramuscular injection every 12 weeks for up to 3 treatments.
  The 80 participants originally treated with topiramate who then received BOTOX® are included in this arm.
- Topiramate: Topiramate starting at a daily oral dose of 25 mg/day titrated up to a maximum dose of 100 mg/day for 36 weeks.
Arm/Group | BOTOX® | Topiramate
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/142
Serious Adverse Events (participants affected / at risk) | 4/220 | 6/142
Other Adverse Events (participants affected / at risk) | 27/220 | 89/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=220) | Topiramate (N=142)
Atrial tachycardia (Cardiac disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=220) | Topiramate (N=142)
Vision blurred (Eye disorders) | 6 | 11
Decreased appetite (Metabolism and nutrition disorders) | 0 | 15
Paraesthesia (Nervous system disorders) | 1 | 44
Dizziness (Nervous system disorders) | 6 | 18
Cognitive Disorder (Nervous system disorders) | 1 | 18
Distubance in attention (Nervous system disorders) | 0 | 12
Sinusitis (Infections and infestations) | 13 | 10
Nausea (Gastrointestinal disorders) | 1 | 19
Fatigue (General disorders) | 1 | 19
Depression (Psychiatric disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT02191579/SAP_000.pdf
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02191579/Prot_001.pdf